CLINICAL TRIAL: NCT04833569
Title: Clinical, Bacterial, and Inflammatory Outcomes of Indocyanine Green-mediated Photodynamic Therapy for Treating Periimplantitis Among Diabetic Patients: a Randomized Controlled Clinical Trial
Brief Title: ICG-PDT, Periimplantitis, Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Labban Nawwaf, Department of Prosthetic Dental Sciences, College of Dentistry, King Saud University, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KingSaud
Record Dates: First submitted 2021-03-30; First posted 2021-04-06 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Peri-Implantitis
Keywords: photodynamic therapy*; periimplantitis*; diabetes mellitus*; indocyanine green*; photosensitizer*
MeSH Terms: conditions — Peri-Implantitis; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Indocyanine green mediated photodynamic therapy (ICG-PDT) (Experimental): Delivery of ICG solution at a concentration of 1 mg/mL will be used. The photosensitizer will be applied until the bottom of the peri-implant pocket using a 1 ml syringe. An 810 nm diode laser (A.R.C. laser GmbH, Nurnberg, Germany) with a power of 200 mW (continuous mode) and total energy of 4 J will be used to excite the ICG by starting from the papilla for 30 s followed by the insertion inside the peri-implant pocket depth for 10 s from both buccal and lingual side moving to coronal direction.
  Interventions: Biological: ICG-PDT; Device: peri-implant mechanical debridement
- Peri-implant mechanical debridement (Placebo Comparator): Non-surgical peri-implant mechanical debridement (PIMD) through ultrasonic device with a carbon tip.
  Interventions: Device: peri-implant mechanical debridement

INTERVENTIONS:
Biological: ICG-PDT — An 810 nm diode laser (A.R.C. laser GmbH, Nurnberg, Germany) with a power of 200 mW (continuous mode) and total energy of 4 J was used to excite the ICG by starting from the papilla for 30 s followed by the insertion inside the peri-implant pocket depth for 10 s from both buccal and lingual side moving to coronal direction. The treatment was applied according to the manufacturer's recommendation. The PDT was performed by a single operator in all test patients
  Arms: Indocyanine green mediated photodynamic therapy (ICG-PDT)
Device: peri-implant mechanical debridement — The peri-implant mechanical debridement was done with the help of ultrasonic carbon tip (Vector, Durr Dental, Bietigheim-Bissingen, Germany).

SUMMARY:
In this study, the effect of photodynamic therapy (indocyanine green mediated) on the clinical, biological and inflammatory aspects was assessed in diabetic patients having peri-implantitis

ELIGIBILITY:
* Inclusion Criteria:

  * adult patients above 45 years of age having type 2 DM
  * HbA1c (≥6.5%) and fasting glucose test
  * probing depth ≥6 mm with bleeding and/or suppuration on at least one site around dental implants that remained in situ
  * On radiographic assessment, the implants exhibited ≥ 3 mm alveolar bone loss apical to the coronal region of the intraosteal portion of the dental implant.
* Exclusion Criteria Patients were excluded if they indicated current or former history of tobacco smoking, any systemic disease other than DM, enrolled in a non-surgical periodontal maintenance program, history of implant repair, pregnancy, and part six months use of antimicrobials, non-steroidal anti-inflammatory drugs, bisphosphonates, or corticosteroids.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2020-09-20 (Actual); Primary Completion 2021-02-15 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Bleeding on probing | 6 months
  Presence or absence of bleeding indicated as '1' or '0', respectively
Plaque index | 6 months
  Presence or absence of plaque indicated as '1' or '0', respectively.
Probing depth | 6 months
  Measurement of consecutive millimeter markings of the periodontal pocket depth
Suppuration | 6 months
  Presence or absence of pus
Crestal bone loss | 6 months
  Measurement of consecutive millimeter markings of the alveolar bone levels

SECONDARY OUTCOMES:
Microbiological analysis (Porphyromonas gingivalis) | 6 months
  Bacterial viability from the peri-implant plaque
Microbiological analysis (Treponema denticola) | 6 months
  Bacterial viability from the peri-implant plaque
HbA1c | 6 months
  Assessment of serum HbA1c
Interleukin-1 beta | 6 months
  Assessment from peri-implant crevicular fluid
Interleukin-6 | 6 months
  Assessment from peri-implant crevicular fluid

CONTACTS AND LOCATIONS:
Overall Officials: Nawwaf Labban, BDS MSD PhD, Principal Investigator — Department of Prosthetic Dental Sciences, College of Dentistry, King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

REFERENCES:
- [Derived] Labban N, Shibani NA, Al-Kattan R, Alfouzan AF, Binrayes A, Assery MK. Clinical, bacterial, and inflammatory outcomes of indocyanine green-mediated photodynamic therapy for treating periimplantitis among diabetic patients: A randomized controlled clinical trial. Photodiagnosis Photodyn Ther. 2021 Sep;35:102350. doi: 10.1016/j.pdpdt.2021.102350. Epub 2021 May 24. PMID 34033934